CLINICAL TRIAL: NCT00878969
Title: Genes, Fibrinolysis and Endothelial Dysfunction- Dialysis Aim 3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment and retention
Sponsor: Vanderbilt University (Other)
Collaborators: University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Fibrinolysis in Dialysis Aim 3; R01HL065193-08A2 (NIH)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Oxidative Stress; Endothelial Dysfunction
Keywords: Hemodialysis; fibrinolysis; oxidative stress; systemic inflammatory reaction; endothelial dysfunction; carotid intima media thickness (IMT; angiotensin receptor blockade; angiotensin converting enzyme inhibition
MeSH Terms: interventions — Valsartan; Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Valsartan (Active Comparator): 80 mg of valsartan (ARB) taken orally on a daily basis for 1 week followed by 160 mg of valsartan taken orally on a daily basis for 18 months
  Interventions: Drug: valsartan (ARB)
- Ramipril (Active Comparator): 2.5 mg of ramipril (ACE inhibitor) taken orally on a daily basis for 1 week followed by 5 mg of ramipril taken orally on a daily basis for 18 months
  Interventions: Drug: ramipril (ACE inhibitor)
- Placebo (Placebo Comparator): matching placebo taken orally on a daily basis for 1 week followed by matching placebo taken orally on a daily basis for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: valsartan (ARB)
  Other Names: Diovan
  Arms: Valsartan
Drug: ramipril (ACE inhibitor)
  Other Names: Altace
  Arms: Ramipril
Drug: Placebo
  Other Names: Inactive pill
  Arms: Placebo

SUMMARY:
The purpose of the study is to see how two classes of blood pressure medications,angiotensin-converting enzyme inhibitors (Ace inhibitors) and angiotensin receptor blockers (ARBs), differ in their long term effects on certain chemicals in the body and on the carotid arteries.

DETAILED DESCRIPTION:
More than 400,000 individuals with chronic kidney disease undergo hemodialysis each year in the United States. Atherosclerotic cardiovascular disease is the leading cause of mortality in these patients. Conventional risk factors for coronary artery disease (CAD) do not adequately explain this increased mortality, whereas biomarker of oxidative stress and inflammation correlate with clinical outcomes. Even with the use of biocompatible membranes, hemodialysis induces a systemic inflammatory reaction characterized by complement activation, leukocyte activation and the generation of reactive oxygen species and cytokines. Oxidative stress and inflammation promote endothelial dysfunction, a predictor of atherosclerotic cardiovascular events.

The purpose of the study is to test the hypothesis that angiotensin-converting enzyme inhibition and angiotensin receptor blockade differ in their long term effects on biomarkers of fibrinolysis, oxidative stress,inflammation and on carotid intima-media thickness (IMT), a predictor of cardiovascular events, in patients with chronic kidney disease undergoing maintenance hemodialysis.

Endogenous Bradykinin (BK) contributes to the hypotensive and pro-fibrinolytic effects of ACE inhibitors. It has been determined that endogenous BK contributes to the vasodilator effects of acute and chronic ACE inhibition. Studies have found that BK stimulates vascular tissue plasminogen activator (t-PA) release through a BK B2 receptor-dependent, nitric oxide (NO) and cyclooxygenase-independent pathway. Hemodialysis patients demonstrates endothelial dysfunction. Data suggests that t-PA release may be attenuated during stimulation of the endogenous kallikrein-kinin system by hemodialysis.

Intra-arterial infusion of BK increases vascular release of F2- isoprostanes, markers of oxidative stress, BK infusions also increase net release of the inflammatory cytokine interleukin-6 (IL-6). Preliminary data raise the possibility that activation of the endogenous kallikrein-kinin system during dialysis could promote inflammation in individuals with chronic kidney disease who are treated with an ACE inhibitor.

Cardiopulmonary bypass activates the endogenous kallikrein-kinin system and causes a systemic inflammatory response. Like hemodialysis, cardiopulmonary bypass activates the endogenous kallikrein-kinin system, increasing BK concentrations. In smokers, who like hemodialysis patients exhibit endothelial dysfunction, the t-PA response to BK was attenuated during cardiopulmonary bypass.

ACE inhibition enhances fibrinolysis and decreases inflammation following cardiopulmonary bypass. The short-term effect of both ACE inhibition and angiotensin II type 1 (AT1) receptors on markers of fibrinolysis and inflammation during dialysis are currently being studied.

Circulating BK concentrations are increased during hemodialysis in individuals treated with an ACE inhibitors compared to those treated with an AT1 receptor blocker.

Bradykinin receptor blockade and the fibrinolytic and inflammatory response to hemodialysis. It is hypothesized that subjects with CAD, the t-PA response to hemodialysis will be blunted compared to that measured in subjects without evidence of CAD, whereas the inflammatory response wil be similar or enhanced.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* On thrice weekly chronic hemodialysis for at least 6 months
* Clinically stable, adequately dialyzed [single-pool Kt/V > 1.2 or Urea Reduction Ratio (URR) > 65%] thrice weekly, with polysulphone membrane for at least 3 consecutive months prior to study

Exclusion Criteria:

* History of functional transplant less than 6 months prior to study
* Use of immunosuppressive drugs within 1 month prior to study
* History of active connective tissue disease
* History of acute infectious disease within one month prior to study
* AIDS (HIV seropositivity is not an exclusion criteria)
* History of myocardial infarction or cerebrovascular event within 3 months
* Advanced liver disease
* Gastrointestinal dysfunction requiring parental nutrition
* Active malignancy excluding basal cell carcinoma of the skin
* History of ACE inhibitor-associated cough (intolerable) or angioedema
* Ejection fraction less than 30%
* Inability to discontinue ACE inhibitor or ARB
* Predialysis potassium repeatedly higher than 6.0 mmol/L (confirmed on a repeated blood draw)
* Anticipated live donor kidney transplant
* Pregnancy or breast-feeding
* History of poor adherence to hemodialysis or medical regimen
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center; Talat A Ikilzer, MD, Principal Investigator — Vanderbilt University Medical Center; Jonathan Himmelfarb, MD, Principal Investigator — University of Washington
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Vanderbilt University Medical Center and at the University of Washington between January 2010 and June 2015.
Pre-assignment Details: There is a 3-week period between enrollment and assignment to treatment group. This "washout" period is to ensure that no blood pressure medicines (ARBs or ACE inhibitors) are left in the body. Although 123 subjects were enrolled, only 78 were assigned to a treatment group (45 subjects were screen failures).
Period: Overall Study
Arm/Group | Valsartan | Ramipril | Placebo
Started | 25 | 27 | 26
Completed | 10 | 12 | 15
Not Completed | 15 | 15 | 11
Not completed — Physician Decision | 5 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 6 | 3
Not completed — kidney transplant | 2 | 3 | 2
Not completed — Adverse Event | 3 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Death | 0 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ramipril: 2.5 mg of ramipril (ACE inhibitor) taken orally on a daily basis for 1 week followed by 6 mg of ramipril taken orally on a daily basis for 18 months
- Total: Total of all reporting groups
Arm/Group | Valsartan | Ramipril | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13) | 53 (13) | 49 (9) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 28
  Male | 14 | 19 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 1 | 10
  Not Hispanic or Latino | 22 | 21 | 25 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 16 | 15 | 44
  White | 10 | 7 | 9 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Interleukin-6 (IL-6)
Description: IL-6 is a sensitive laboratory assay for serum levels of interleukin-6, which is a pro-inflammatory cytokine used to evaluate the inflammatory response.
Time Frame: baseline and 18 months
Population: Based on our power calculations, we needed 210 subjects to complete the study to be able to detect an effect. Given that only 37 subjects completed the study (18% of goal), no formal analyses were performed. Specifically, data were not collected for this assessment for any of the participants enrolled in the study.
Arm/Group | Valsartan | Ramipril | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Valsartan | Ramipril | Placebo
Serious Adverse Events (participants affected / at risk) | 8/25 | 9/27 | 9/26
Other Adverse Events (participants affected / at risk) | 19/25 | 15/27 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valsartan (N=25) | Ramipril (N=27) | Placebo (N=26)
infection (Infections and infestations) | 1 (1) | 3 (5) | 2 (3)
pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (2)
cardiac (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
electroyte disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (3)
hypertension/hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (3)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0)
GI upset (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
generalized symptoms (General disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2)
access related (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
trauma (General disorders) | 1 (1) | 0 (0) | 0 (0)
pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
blood clot (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
suicide ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
excessive bleeding (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
excessive fluid in abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valsartan (N=25) | Ramipril (N=27) | Placebo (N=26)
access related (Vascular disorders) | 8 (12) | 5 (15) | 5 (17)
GI upset (Gastrointestinal disorders) | 2 (4) | 5 (8) | 8 (16)
cardiac (Cardiac disorders) | 4 (7) | 5 (7) | 5 (7)
neurological (Nervous system disorders) | 2 (3) | 2 (11) | 2 (5)
hypertension/hypotension (Vascular disorders) | 6 (6) | 7 (9) | 0 (0)
electrolyte disorder (Metabolism and nutrition disorders) | 2 (10) | 3 (3) | 2 (2)
pain (General disorders) | 3 (4) | 2 (2) | 4 (8)
pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 3 (3)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 4 (4)
infection (Infections and infestations) | 4 (4) | 0 (0) | 3 (4)
generalized symptoms (General disorders) | 2 (2) | 5 (6) | 0 (0)
trauma (General disorders) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes